CLINICAL TRIAL: NCT03183323
Title: Implementation of Telerehabilitation In Support of HOme-based Physical Exercise for Heart Failure
Acronym: ITISHOPE4HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LH2017_HOPE4HF
Record Dates: First submitted 2017-05-30; First posted 2017-06-12 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure, Systolic; Heart Failure, Diastolic; Chronic Kidney Diseases; Cardiorenal Syndrome
Keywords: hfpef; hfref; cardiorenal syndrome; exercise; telerehabilitation; rehabilitation
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure, Diastolic; Renal Insufficiency, Chronic; Cardio-Renal Syndrome; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: RCT, 1:1 into telerehabilitation or standard care. Patients will be stratified by EF >/< 40 %, age >/< 60 years and by sex.
Who Masked: Outcomes Assessor
Masking Description: Group assignment is not masked at performance tests. Group assignment is masked to the echo/MRI technician, and for investigators interpreting the recordings.
  Masking is not relevant for laboratory analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): In addition to optimal medical treatment: 3 months of twice weekly group-based telerehabilitation through a video-conferencing on a tablet platform. In addition access to instruction videos for further self-training through the same platform and throughout the whole 2-year period. Electronic devices to trace activity.
  Interventions: Behavioral: Telerehabilitation
- Standard care (No Intervention): In addition to optimal medical treatment: Advice on physical activity. Electronic devices to trace activity.

INTERVENTIONS:
Behavioral: Telerehabilitation — Activity trackers. Mio Slice is worn through the whole study. Actigraph is worn for one week, at 4 different timepoints through the study.
  Other Names: Mio Slice; Actigraph
  Arms: Telerehabilitation

SUMMARY:
ITISHOPE4HF is a randomized controlled trial of telerehabilitation in a heart failure population. The goal is to evaluate if a home-based telerehabilitation project can increase physical activity in heart failure patients. Patients will be provided telerehabilitation or advice on physical activity (standard care).

DETAILED DESCRIPTION:
Outpatient cardiac rehabilitation programs are well documented as an important part of treatment and care for heart failure patients. Training with instruction gives the participant a commitment to participate. The result is increased activity compared to controls.

This trial will include participants from the about 75 % of heart failure patients who for some reason do not participate in regular outpatient rehabilitation. Distance to rehabilitation centers and the psychological burden of a group setting are believed to be important reasons for not participating. Telerehabilitation can hopefully overcome these hurdles for many patients, and thereby provide instructed training for these patients.

The trial will also include patients with renal disease. Heart disease is the main cause of death in patients with renal disease, even at younger ages. Because of the complexity of both optimal medical treatment and fluid balance, these patients are often not included in clinical trials. The cardiorenal crosstalk will be explored, how in influence the heart failure phenotypes and the response to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure (HFpEF or HFrEF) according to European guidelines.
* Moderate or severe signs and symptoms of heart failure (NYHA II-III) in the 6 months prior to enrolment.
* N-terminal pro brain natriuretic peptide (NT-proBNP) > 300 pmol/L.
* Stable (> 4 weeks) medical therapy for risk factor control.
* Capability to provide signed, informed, written consent.

Exclusion Criteria:

* Attendance at a rehabilitation program in the 6 months prior to enrolment.
* Non-heart failure causes of heart failure symptoms (significant valvular disease, coronary disease available for revascularization, uncontrolled hypertension, arrhythmia).
* severe or very severe pulmonary disease (eg. COPD GOLD III-IV).
* presence of conditions which might prevent patients from safely exercising at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Improvement in long-term physical activity. | 2 years
  Change in physical activity between intervention and control group measured throughout the study with Actigraph activity trackers from baseline to 2 years.

SECONDARY OUTCOMES:
Changes in cardiac structure and function. | 2 years.
  Echocardiographic indices - improvements from exercise.
Change in physical fitness. | 2 years
  The change in physical fitness at from baseline to 2 years follow-up.
Effects on renal function. | 2 years.
  Changes in renal function (GFR/proteinuria) by exercise.
Long-term effects on cardiovascular risk factors. | 2 years.
  Blood measurements of Cardiac risk factors.
Effects on endothelial function. | 2 years.
  Changes in peripheral arteries measured by vascular ultrasound from baseline to two years follow-up..
Change in long-term quality of life. | 2 years.
  Measured via validated questionnaires at different point during follow-up.
Mid-term morbidity | 2 years
  Evaluate morbidity as hospitalization of cardiovascular causes
Mid-term mortality | 2 years
  Mortality during follow-up

OTHER OUTCOMES:
Differences in heart failure presentation associated with co-morbid chronic kidney disease. | Baseline.
  Evaluated by cardiac imaging.
The association of cardiac fibrosis with cardiorenal syndrome | Baseline
  Evaluated by echo cardiography and/or cardiac MRI including T1 mapping.
Feasibility of telerehabilitation | 6 months.
  Assessment of the proportion of completed telerehabilitation programs
Validation of the Mio Slice as a scientific activity tracker. | 6 months
  Comparison of data from the Mio Slice with reference to validate it as a scientific tool for monitoring heart failure patients
Urine metabolomics Associated With heart failure phenotypes. | Baseline.
  Comparing traits in urine metabolomics between participants with and without chronic kidney disease. Comparing with earlier studies of patients with chronic kidney disease and healthy controls.
Long-term changes in urine metabolomics after intervention. | 2 years.
  Looking for changes in metabolomics expression caused by exercise.
Cost-effectiveness of telerehabilitation | 1 years.
  Vs. outpatient rehabilitation
Change in physical fitness | 6 months
  Evaluate short-term effect of telerehabilitation on measurements of physical fitness
The influence of cardiorenal characteristics on training effect | 6 months
  Evaluate if cardiorenal characteristics influence on change in peak oxygen consumption of training
Do renal function modulate the training effect on cardiac remodeling | 12 months
  Evaluate if renal function modulate the training effect on changes in cardiac characteristics
Change in short-term quality of life. | 6 months
  Patient reported outcomes after training intervention

CONTACTS AND LOCATIONS:
Overall Officials: Havard Dalen, MD, PhD, Principal Investigator — Norwegian University of Science and Tehnology
Locations (1):
- St. Olav University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Will follow the regulations and policy decided by the Norwegian University of Science and Technology

REFERENCES:
- [Derived] Lundgren KM, Langlo KAR, Salvesen O, Aspvik NP, Mo R, Ellingsen O, Vesterbekkmo E, Zanaboni P, Dalen H, Aksetoy IA. Exercise-Based Telerehabilitation for Heart Failure Patients Declining Outpatient Rehabilitation-A Randomized Controlled Trial. Med Sci Sports Exerc. 2025 Mar 1;57(3):449-460. doi: 10.1249/MSS.0000000000003590. Epub 2024 Nov 6. PMID 39501477
- [Derived] Lundgren KM, Langlo KAR, Salvesen O, Zanaboni P, Cittanti E, Mo R, Ellingsen O, Dalen H, Aksetoy IA. Feasibility of telerehabilitation for heart failure patients inaccessible for outpatient rehabilitation. ESC Heart Fail. 2023 Aug;10(4):2406-2417. doi: 10.1002/ehf2.14405. Epub 2023 May 23. PMID 37221704